CLINICAL TRIAL: NCT02420093
Title: Investigating the Clinical Effects of Supporting Neutral Pelvic Position in Sitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oakland University (Other)
Responsible Party: Principal Investigator, Patricia Connors, Patricia Connors - Doctoral Student, Oakland University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRBnet # 679149-4
Record Dates: First submitted 2015-01-23; First posted 2015-04-17 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2016-11

CONDITIONS: Low Back Pain; Strain; Postural
MeSH Terms: conditions — Low Back Pain; Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): The experimental group will use the "Pelvis Support Assembly" per US Patent number US 8,857,906 B2, in the seat of their work or home desk chairs as tolerated during the 3 weeks intervention interval. This pelvic support device supports the user from the pelvis and aids in maintaining a more anatomically neutral lumbar and pelvic position in sitting.
  Interventions: Device: "Pelvis Support Assembly"
- Control Group (No Intervention): The control group will not use the "Pelvis Support Assembly" per US Patent number US 8,857,906 B2 but will continue in their current sitting arrangement during the same 3 week interval

INTERVENTIONS:
Device: "Pelvis Support Assembly" — Use of a portable and adjustable "Pelvis Support Assembly" in the seat of the subject's work or home desk chairs as tolerated during the 3 weeks intervention interval. This pelvic support device supports the user from the pelvis and aids in maintaining a more anatomically neutral lumbar and pelvic position in sitting. This device is not officially named at this time but is as represented in US Patent number is US 8,857,906 B2.
  Arms: Experimental Group

SUMMARY:
The aim of this study is to examine the clinical effects of supporting the human pelvis in a neutral sitting position in subjects with Low Back Pain over a 3-week period. The neutral sitting posture will be supported by a portable and adjustable "pelvic support device" or "pelvic support assembly" per US Patent number US 8,857,906 B2 that is used in the seat of the user's desk chair.

DETAILED DESCRIPTION:
This study is a randomized control trial with repeated measures. It will include 34 subjects with low back pain who sit 25 hours a week or more at a desk / computer.

There will be 2 groups: control and experimental, each with 17 subjects. All subjects will be measured on the same 2 dates (3 weeks apart - pre and post intervention) with the same measures.

The experimental group will use a pelvic support device, that aids in supporting the user's pelvis in a neutral position, in their desk chairs at home or work as tolerated during this 3 weeks.

The control group will continue in their current sitting arrangement during the same 3 weeks.

For control of conflict of interest, the Sponsor-Investigator will not perform any of the measures and data will be coded for subject group assignment until all data analysis is finalized.

Multiple sessions of 3-week intervals of data collection may be performed as needed to achieve desired subject number in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a history of 1 or more episodes of low back pain (LBP) in the last calendar year or who currently has LBP without radiation of pain from the low back into the legs.
2. Males or Females who are 20-65 years of age.
3. Individuals who engage in work that requires sitting at a desk or computer 25 or more hours a week.
4. Individuals who plan to work full time for each of the 3 weeks of the trial (April. 22 - May. 14, 2015), with no planned business travel or time off.
5. Individuals who can commit to attending two 1-1.5 hours data collection events (appointments times from 4:30-8:30 pm): Either on: Wed. April 22, 2015 and Wed May 13, 2015 or Thurs. April 23, 2015 and Thurs. May 14, 2015 at a location on the west side of Ann Arbor, MI.
6. Individuals who can read, write and understand English fluently. (Questionnaires are in English)
7. Individuals who, while maintaining upright sitting, can lift their knee approximately 3-6 inches off the chair (as in marching), one at a time, on both sides.
8. Individuals who are willing to wear non-binding or flexible clothing around their hips and pelvis at work during the three weeks of the trial if chosen to be in the experimental group. Note: Because the posture device being studied tilts the user's pelvis more upright, compared to the common slump / backward pelvic tilt that occurs in sitting, some find, especially males , that this binds them in the front of their pelvis and groin area when their clothing is tight or restrictive. Looser or flexible clothing has significantly aided in tolerance of this positioning and will be recommended if subject is chosen to be in the experimental group, assigned to use the device.

Exclusion Criteria:

1. Individuals who currently have pain radiating from low back into the legs below hips.
2. Individuals with a history of low back surgery that includes:

   * Spinal Fusion at any level
   * Placement of any plates or screws in the low back (Note: those with a history of back surgery > 1 year ago that did not involve plates or screws and are not under medical restrictions associated with their back will be accepted.)
3. Individuals who have had any kind of lumbar surgery within the last calendar year.
4. Individuals with a currently painful coccyx area or a history of broken coccyx (or tailbone) less than 1 year ago.
5. Individuals with a history of total hip replacement in the last year.
6. Individuals with significantly limited and painful back backward bending.
7. Anyone with known lumbar anterolisthesis (or forward slippage of 1 vertebra on another) > grade 1
8. Anyone believing they may be more than 2 months pregnant at the time of the study.
9. Anyone who is not able to lie on their stomach for any reason.
10. Anything not listed above but known to subject that makes them believe they will be unable to meet the requirements of the study as outlined.

    -

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Connors, MSPT, Principal Investigator — Oakland University Doctoral Student; Melodie Kondratek, MS, DScPT, Study Chair — Oakland University
Locations (1):
- Gladwin Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 9 | 8
Completed | 8 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Oswestry Low Back Pain Disability Index
Description: This questionnaire measures the impact subject's low back pain on functional tolerance levels. Scale range is 0-100 with the lower score indicating a higher functional / activity level as it relates to Low Back Pain.
Time Frame: Baseline and 3 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 8 | 7
units on a scale | -8.25 (1.62) | -0.86 (1.43)

2. Primary Outcome: Change in Left and Right Hamstring Length Testing
Description: This test measures left and right hamstring length of the subject while they are lying on their back. The angle between the femur and tibia/fibula were measured when the hip angle held constant at 90 degrees and knee in full amount of available knee extension. This measure will use inclinometers for measurement.
Time Frame: Baseline and 3 Weeks
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 8 | 7
degrees
  Left Hamstring | 4.79 (4.95) | 0.19 (1.89)
  Right Hamstring | 1.71 (4.41) | 2.38 (3.06)

3. Primary Outcome: Change in Sorenson Test for Lumbar Muscle Endurance
Description: This test measures a persons back strength in 1 repetition of holding a back posture in neutral as long as can while lying on their stomach, legs stabilized on a treatment table.
Time Frame: Baseline and 3 Weeks
Measure: Mean (Standard Deviation); unit: time in seconds
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 8 | 7
time in seconds | 5.88 (2.19) | 4.07 (2.68)

4. Primary Outcome: Change in Fingertip to Floor Flexibility Test
Description: This test measures subjects flexibility in forward trunk bending while subject is standing on a block 20 cm high. Measurement is in centimeters from fingertip to edge of step, above or below the step edge.
Time Frame: Baseline and 3 Weeks
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 8 | 7
centimeters | 1.25 (0.94) | 0.71 (1.60)

5. Primary Outcome: Change in Numeric Pain Rating Scale
Description: This questionnaire measures subjective perception of pain levels on a 0-10 (11 point) scale, with "0" being "no pain" and "10" being the "worst pain imaginable".
Time Frame: Change from Baseline after 3 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 8 | 7
units on a scale | -1.5 (0.433) | -0.18 (0.34)

ADVERSE EVENTS:
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No